CLINICAL TRIAL: NCT05162690
Title: Efficacy of Dapagliflozin in Diabetes Associated Peripheral Neuropathy: A Randomized Placebo Controlled Trial
Brief Title: Efficacy of Dapagliflozin in Diabetes Associated Peripheral Neuropathy
Acronym: DINE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGIMER1
Record Dates: First submitted 2021-10-27; First posted 2021-12-17 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; SGLT2 inhibitors; dapagliflozin; CCM; IENFD; Skin Biopsy; Peripheral Neuropathy; Corneal confocal microscopy; intraepithelial nerve fiber density; Diabetic Sensory Polyneuropathy(DSPN); DSPN
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Drug Arm (Active Comparator): Dapagliflozin 10 milligram Once a day
  1 year
  Interventions: Drug: Dapagliflozin 10 milligram
- The Placebo Arm (Placebo Comparator): Metformin 1gram Per Oral Twice a day Glimepiride 2 milligram oral twice a day Dipeptidyl peptidase 4 inhibitors (DPP4 inhibitors)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 milligram — 10mg per day of Dapagliflozin will be given to the patients
  Arms: The Drug Arm
Other: Placebo — Metformin DPP4 inhibitors
  Arms: The Placebo Arm

SUMMARY:
Diabetic peripheral neuropathy(DPN) is a length dependent axonal neuropathy that affects at least 50% of patients with diabetes mellitus. DPN is often asymptomatic during the early stages of diabetes ,however, once symptoms and overt deficits have developed, it cannot be reversed. Early diagnosis of neuropathy is important because early diagnosis and timely intervention might prevent the development and progression of diabetic neuropathy.Though glycemic control has been shown to prevent the progression of diabetic microvascular complications including diabetic peripheral neuropathy in Type I DM, such strict glycemic control has not shown to improve diabetic peripheral neuropathy in Type 2 DM. There are only few animal studies conducted so far which have shown that the use of SGLT2 inhibitors prevents the progression of diabetic peripheral neuropathy.Thus the investigators postulate that the use of SGLT2 inhibitor in patients with Type 2 Diabetes Mellitus might be beneficial in the prevention of progression of diabetic peripheral neuropathy as well as reverse it.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy is a length dependent axonal neuropathy that affects at least 50% of patients with diabetes mellitus. It is characterized by sensory loss and pain that initially affects small unmyelinated C fibers which is followed by involvement of the large myelinated fibers as diabetes progresses. DPN is often asymptomatic during the early stages of diabetes ,however, once symptoms and overt deficits have developed, it cannot be reversed. Early diagnosis of neuropathy is thus important because early diagnosis and timely intervention might prevent the development and progression if diabetic neuropathy and might provide us with a means to identify patients at high risk for future complications of DPN which includes risk of foot ulcers and lower limb amputation.

Methods to quantify neuropathy include clinical scores based on symptoms and neurological tests, quantitative sensory testing, electrophysiological measurements, in the form of nerve conduction studies and intraepidermal nerve fiber density in skin biopsy specimens. The neurological examination involves an assessment, such as modified neuropathy disability score, a composite score that assesses touch, temperature and vibration perception and reflexes, which require expert clinical judgement, a strong element of subjectivity and hence poor reproducibility. Neurophysiology is objective and reproducible and is currently considered to be the most reliable measurements for confirming the diagnosis of diabetic neuropathy. However, these measures mainly assess large nerve fibers, making them less sensitive to early DPN,which is more likely to involve the small fibers to begin with.

Objective measures are thus required to accurately determine nerve pathology to detect early stages of DPN, which may be more susceptible to intervention than late-stage sequelae. Small ﬁbers, which constitute 70-90% of peripheral nerve ﬁber, may be measured in skin biopsies by assessing intraepidermal nerve ﬁber density, which is considered to be the gold standard for the evaluation of small fibers damage. Indeed, the European Federation of the Neurological Societies and the Peripheral Nerve Society endorse intraepidermal nerve fiber quantification to confirm the clinical diagnosis of small fiber neuropathy with a strong (Level A)recommendation.

Recently, corneal confocal microscopy (CCM), a noninvasive modality for the study of the human cornea, has emerged as a promising technique for the detection of small nerve ﬁber alterations. CCM is a rapid non-invasive imaging technique for the quantitative assessment of small fiber damage. Several studies have shown that it has good diagnostic utility for sub-clinical DPN, predicts incident DPN and correlates with other measures of neuropathy . Furthermore, automated quantification of corneal nerve parameters allows rapid, unbiased and objective assessment of small fiber damage with comparable diagnostic capability to intraepithelial nerve fiber density (IENFD). Recent data also suggest that CCM shows good reproducibility and could be useful to document nerve regeneration after treatment and simultaneous pancreas and kidney transplantation.

There is currently no Food and Drug Administration (FDA) approved therapy to prevent or reverse human DPN. The current management approach focuses on reasonable glycemic control, and management of associated pain. Sodium-glucose cotransporter 2 (SGLT2) inhibitors as oral hypoglycemic agents have been approved for treating type 2 diabetes mellitus (T2DM). The insulin-independent action mechanism and extra-metabolic benefits of these agents have encouraged ongoing preclinical and clinical trials for evaluating the efficacy and safety of SGLT2 inhibitors. In addition to glucose-lowering effects without hypoglycemia, SGLT2 inhibitors retard the development and progression of diabetic complications. However, it is uncertain whether this effect of SGLT2 inhibitors is due to their glucose-lowering effect or not. In addition, unlike diabetic nephropathy, the effects of SGLT2 inhibitors on diabetic peripheral neuropathy are unexplored.

To date, only three studies regarding the effects of SGLT2 inhibitors for DPN in T2DM animal models are reported. Investigators evaluated neuronal effects in terms of simple functional parameters, such as motor nerve conduction velocity and tail flick test. Results of these studies verified the beneficial effects of SGLT2 inhibitors for DPN, and these effects were considered to indirect effects of the improvement of hyperglycemia.

Since no human studies have yet been conducted using SGLT2 inhibitors in the prevention and progression of diabetic neuropathy, hence, investigators plan to conduct a randomized controlled trial evaluating the efficacy of dapagliflozin in diabetic peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

-

Type 2 Diabetes Mellitus < 5 years duration

Age >18yrs

Presence of neuropathy at baseline (accessed by Michigan Neuropathy Screening Instrument score >7 )

estimated Glomerular Filtration rate (eGFR) > 45ml/min/m2

HBA1c < 9

Exclusion Criteria:

Untreated Hypothyroidism

Patients currently on SGLT2 inhibitors History of Leprosy

Patients with history of and current foot ulcers

Presence of Peripheral Vascular disease(ABI <0.9)

B12(<200 pg/ml)/ Folate (<4.6 ng/ml)

History of alcohol abuse (>2 standard drink per day for males and >1 standard drink for females)

Factors affecting corneal nerves( severe dry eyes, severe corneal dystrophies, ocular trauma or surgery in the preceding 6 months)

Negative consent

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraepithelial nerve fiber density | 24 weeks
  mean change in intraepithelial nerve fiber density(F/mm) will be evaluate at baseline and after 24 weeks of treatment with dapagliflozin.

SECONDARY OUTCOMES:
corneal nerve fiber density | 24 weeks
  mean change in corneal nerve fiber density (total number of nerves per square millimeter of corneal tissue) will be evaluated at baseline and after 24 weeks of treatment with dapagliflozin.

CONTACTS AND LOCATIONS:
Overall Officials: Ashu Rastogi, DM, Principal Investigator — PGIMER, India
Locations (1):
- Department of Endocrinology, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adhikari U, Gad H, Chatterjee D, Malhotra C, Bhadada SK, Malik RA, Rastogi A. Dapagliflozin for Small Nerve Fibre Regeneration in Diabetic Peripheral Neuropathy: A Randomised Controlled Study (DINE). J Peripher Nerv Syst. 2025 Mar;30(1):e70011. doi: 10.1111/jns.70011. PMID 40044634